CLINICAL TRIAL: NCT00383812
Title: Intravitreal Bevacizumab for Polypoidal Choroidal Vasculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bevacizumab for PCV
Record Dates: First submitted 2006-10-03; First posted 2006-10-04 (Estimated); Last update posted 2006-10-04 (Estimated); Status verified 2006-10

CONDITIONS: Polypoidal Choroidal Vasculopathy
Keywords: Polypoidal choroidal vasculopathy; Intravitreal Bevacizumab
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy

INTERVENTIONS:
Drug: Intravitreal Bevacizumab

SUMMARY:
1. Primary objectives

   a. To evaluate the Effects of intravitreal Bevacizumab on polypoidal choroidal vasculopathy(PCV)
2. Secondary objectives

   1. To assess the changes in visual acuity
   2. To assess the change in lesion characteristics of PCV

      * size of PCV
      * fluorescein leakage
      * foveal thickness
   3. To investigate the safety of intravitreal Bevacizumab in patients with PCV
   4. To assess the effect of intravitreal Bevacizumab on the recurrence rate and the the incidence of submacular hemorrhage in patients with PCV

ELIGIBILITY:
Inclusion Criteria:

* Male or female, CNV secondary to PCV
* BCVA of 20/40 to 20/320 (Snellen equivalent)
* Evidence of presumed recent disease progression (blood, growth by FA, or recent VA loss)

Exclusion Criteria:

* Uncontrolled glaucoma or any other ocular condition that would prevent an improvement in visual acuity
* Media opacity in the study eye that precludes clinical and photographic evaluation
* Intraocular surgery < 1 month before day 0
* Use of heparin/warfarin within 1 month prior to injection
* Known allergy or hypersensitivity to fluorescein, indocyanine green or povidone iodine
* Contraindication to pupil dilation in either eye
* Any condition which precludes patients' ability to comply with study requirements including completion of the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-05; Study Completion 2008-05

PRIMARY OUTCOMES:
To assess the percentage of patients who gained an improvement in best corrected visual acuity (BCVA) by 15 letters of more.
To assess the percentage of patients whose final visual acuity resulted in Snellen equivalent of 20/200 or worse

SECONDARY OUTCOMES:
To investigate the resolution time of macular edema, subretinal fluid, and/or pigment epithelial detachment (PED) using optical coherence tomography (OCT)
To evaluate change in size and leakage of PCV, using fluorescein angiography (FA) and/or indocyanine angiography (ICGA)

CONTACTS AND LOCATIONS:
Overall Officials: Young Hee Yoon, MD, Principal Investigator — Asan Medical Center; June-Gone Kim, MD, Principal Investigator — Asan Medical Center; Sun Young Lee, MD, Principal Investigator — Asan Medical Center; Hyewon Chung, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea